CLINICAL TRIAL: NCT03891342
Title: Comparing of Two Regimes (Fast and Slow) of Fluid Challenge on Glycocalyx Assessed by Perfused Boundary Region in Septic and Elective Major Surgical Patients
Brief Title: Effect of Fluid Challenge on Glycocalyx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Hradec Kralove (Other)
Collaborators: University Hospital Pilsen (Other)
Responsible Party: Principal Investigator, Vladimir Cerny, Principal Investigator, University Hospital Hradec Kralove
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AZVCR 9307_1
Record Dates: First submitted 2017-10-24; First posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Anesthesia; Endothelial Dysfunction; Sepsis; Septic Shock; Surgery
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with sepsis/septic shock (Experimental): Comaprison of fast or slow fluid bolus administration in patients with sepsis/septic shock 48hours before admission to ICU requiring fluid challenge as assessed by clinical examination
  Interventions: Drug: Fluid bolus administration
- Major surgical patients (Experimental): Comaprison of fast or slow fluid bolus administration in patients undergoing major surgery requiring fluid challenge as assessed by clinical examination
  Interventions: Drug: Fluid bolus administration

INTERVENTIONS:
Drug: Fluid bolus administration — Fluid bolus administration either "fast" in 5 minutes or "slow" in 30minutes.
  Other Names: Fluid challenge

SUMMARY:
Interventional study comparing effect of two regimes of fluid challenge in patients with sepsis and in patients undergoing elective major surgery on glycocalyx by using perfused Boundary Region in sublingual microcirculation.

DETAILED DESCRIPTION:
Effect of two regimes of fluid challenge on GCX in patients with sepsis and during elective surgery under general anesthesia.

Hypothesis to be tested: Administration of 500 ml of balanced solution as a bolus impairs GCX more than prolonged administration.

The aim of the study: Comparison of two regimes of fluid challenge in patients with sepsis and in patients undergoing elective major surgery.

Type of the study: Open, randomized, interventional.

Subjects:

Part A: Patients with sepsis within 48 hours before admission to ICU requiring fluid challenge based on clinical or echocardiographic assessment.

Part B: Patients during major elective surgery requiring fluid challenge based on clinical or echocardiographic assessment.

Sample size calculation (based on expected difference in PRB, alpha error I =0,05 and study power = 0,99) = 52 patients. Investigators plan enrolment of 60 patients for each part, totally 120 patients.

Intervention:

* 500 ml of balanced crystalloid solution within 5 minutes (group "fast")
* 500 ml of balanced crystalloid solution within 30 minutes (group "slow") Data to be recorded and analysed: Demographics, severity score, fluid response assessment, sublingual microcirculation by SDF imaging will be recorded at time points: baseline, after intervention, after 60 minutes, after 120 minutes, plasma syndecan-1 will be analysed before intervention and 120 minutes thereafter, microcirculatory data and Perfused Boundary Region.

ELIGIBILITY:
Inclusion Criteria:

arm A: age over 18, diagnosis sepsis, fluid bolus administration indicated, arm B: age 18-70, ASA status I-III, major surgery

Exclusion Criteria:

none.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Influence of balanced crystalloid infusion time on endothelial glycocalyx | baseline and at 20, 40, 60 and 120 minutes
  Change in the endothelial glycocalyx thickness by PBR method

CONTACTS AND LOCATIONS:
Overall Officials: Jan Benes, Assoc.Prof., Principal Investigator — Charles University hospital in Plzen, Czech Republic
Locations (1):
- FN Plzen, Pilsen, Czechia

IPD SHARING:
Plan to Share IPD: Undecided